CLINICAL TRIAL: NCT00511238
Title: An Open-label, Single-arm, Phase 2 Study of Carfilzomib in Patients With Relapsed and Refractory Multiple Myeloma
Brief Title: Phase 2 Study of Carfilzomib in Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PX-171-003
Record Dates: First submitted 2007-08-01; First posted 2007-08-03 (Estimated); Results first posted 2013-12-09 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Multiple Myeloma
Keywords: Onyx; PR171; carfilzomib; multiple myeloma; relapsed; refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — carfilzomib; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- carfilzomib (A0) (Experimental)
  Interventions: Drug: carfilzomib
- carfilzomib (A1) (Experimental)
  Interventions: Drug: carfilzomib

INTERVENTIONS:
Drug: carfilzomib — Subjects will receive carfilzomib 20 mg/m2 as an intravenous bolus over 2 minutes on Days 1, 2, 8, 9, 15, and 16 of 28 day cycles. A maximum of 12 cycles will be administered.
  Other Names: PR-171; PR171; Kyprolis® (carfilzomib) for Injection
  Arms: carfilzomib (A0)
Drug: carfilzomib — Subjects will receive carfilzomib intravenously over up to 10 minutes on Days 1, 2, 8, 9, 15, and 16 of 28 day cycles. In cycle 1, the dose is 20 mg/m2. If all doses are administered and well-tolerated over Cycle 1, beginning with Cycle 2 the dose will escalate to 27 mg/m2 cycle. A maximum of 12 cycles will be administered.
  Other Names: PR-171; PR171; Kyprolis® (carfilzomib) for Injection
  Arms: carfilzomib (A1)

SUMMARY:
To evaluate the overall response rate and safety and tolerability of carfilzomib in subjects with relapsed and refractory multiple myeloma.

Patients must have received prior treatment with bortezomib and either thalidomide or lenalidomide and be refractory to their last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Disease Related

  * Multiple myeloma
  * Subjects must have measurable disease defined as one of the following:

    * Serum M-protein ≥ 1 g/dL
    * Urine M-protein ≥ 200 mg/24 hours
    * Serum FLC ≥ 10 mg/dL with abnormal ratio (A0 Only)
    * Quantitative immunoglobulin levels using nephelometry or turbidometry (only if protein electrophoresis was felt to be unreliable for M-protein measurement) (A0 Only)
  * Subjects must have been responsive (i.e., achieved an MR or better) to first-line, standard of care therapy
  * Refractory to the most recently received therapy. Refractory disease is defined as ≤ 25% response or progression during therapy or within 60 days after completion of therapy.
  * Subjects must have received ≥ 2 prior regimens for relapsed disease. Induction therapy and stem cell transplant will be considered as one regimen (A1 Only)
  * Subjects must have received prior treatment with bortezomib, and either thalidomide or lenalidomide
  * Subjects must have received an alkylating agent either alone or in combination with other myeloma treatments (history of stem cell transplant is acceptable) (A1 Only)
  * Subjects must have received an anthracycline either alone or in combination with other myeloma treatments, unless not clinically indicated (A1 Only)
* Demographic

  * Males and females > 18 years of age
  * Life expectancy of more than three months
  * Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Laboratory

  * Adequate hepatic function, with bilirubin less than 2.0 times the upper limit of normal, and AST and ALT of less than 3.0 times the upper limit of normal
  * Uric acid within normal range (A0 Only)
  * Total white blood cell (WBC) count ≥ 2.0 × 109/L, absolute neutrophil count (ANC) ≥ 1.0 × 109/L, hemoglobin ≥ 8.0 g/dL, and platelet count ≥ 50.0 × 109/L (A0 Only)
  * Absolute neutrophil count > 1,000/mm3, hemoglobin > 8.0 g/dL, and platelet count > 50,000/mm3 (A1 Only)

    * Subjects should be platelet transfusion independent
    * Screening ANC should be independent of G-CSF or GM-CSF support for ≥ 1 week and of pegylated G-CSF for ≥ 2 weeks
    * Subjects may receive red blood cell (RBC) or platelet transfusions or receive supportive care such as erythropoietin and darbepoetin in accordance with institutional guidelines
  * Calculated and measured creatinine clearance of ≥ 30 mL/minute, calculated using the formula of Cockcroft and Gault [(140 - Age) X Mass (kg) / (72 X Creatinine mg/dL)]. Multiply result by 0.85 if female.
* Ethical / Other

  * Written informed consent in accordance with federal, local, and institutional guidelines
  * Female subjects of child-bearing potential must have a negative serum pregnancy test within seven days of the first dose and agree to use dual methods of contraception during and for 3 months following last dose of drug. Post menopausal females (> 45 years old and without menses for > 1 year) and surgically sterilized females are exempt from a pregnancy test. Male subjects must use an effective barrier method of contraception during study and for 3 months following the last dose if sexually active with a female of child-bearing potential.

Exclusion Criteria:

* Disease Related

  * Multiple Myeloma IgM (A1 Only)
  * Subjects who failed to achieve at least a confirmed MR(≥ 25% reduction in M-protein for ≥ 6 weeks) (A1 Only)
  * Subjects with non-secretory multiple myeloma, defined as < 1 g/dL M-protein in serum and < 200 mg/24 hr M-protein in urine
  * Subjects with disease measurable only by serum free light chain (SFLC) analysis (A1 Only)
  * Glucocorticoid therapy (prednisone > 10 mg/day orally or equivalent) within the last three weeks
  * POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
  * Plasma cell leukemia
  * Chemotherapy with approved or investigative anticancer therapeutics including steroid therapy within the three weeks prior to first dose
  * Radiation therapy or immunotherapy in the previous four weeks; localized radiation therapy within 1 week prior to first dose
  * Participation in an investigational therapeutic study within three weeks or within five drug half-lives (t1/2) prior to Day 1, whichever time is greater
  * Prior treatment with carfilzomib
* Concurrent Conditions

  * Major surgery within three weeks before Day 1
  * Congestive heart failure (New York Heart Association class III to IV), symptomatic cardiac ischemia, cardiomyopathy, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction in the previous six months, LVEF < 40
  * Acute active infection requiring systemic antibiotics, antivirals or antifungals within 2 weeks prior to first dose
  * Known or suspected HIV infection or subjects who are HIV seropositive
  * Active hepatitis A,B,or C infection
  * Non-hematologic malignancy within the past three years except a) adequately treated basal cell or squamous cell skin cancer, b) carcinoma in situ of the cervix, or c) prostate cancer <Gleason Grade 6 with stable PSA
  * Subjects with treatment related myelodysplastic syndrome
  * Significant neuropathy (Grade 3, 4 or Grade 2 with pain) at the time of study initiation
  * Subjects in whom the required program of oral and intravenous fluid hydration is contraindicated, e.g., due to pre-existing pulmonary, cardiac or renal impairment (A1 Only)
  * Subjects with known or suspected amyloidosis (A1 Only)
  * Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis (A1 Only)
  * Any clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent (A1 Only)
* Ethical / Other

  * Female subjects who are pregnant or lactating
  * Serious psychiatric or medical conditions that could interfere with treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2007-08; Primary Completion 2010-11 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (34):
- United States (28):
  - Southern Cancer Center, Mobile, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope National Medical Center, Duarte, California
  - Scripps Clinic, La Jolla, California
  - University of California, San Francisco, San Francisco, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Northwestern Universtiy, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - St. Vincent Catholic Medical Center, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Oncology & Hematology Care, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Northwest Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Cross Cancer Institute, Edmonton, Alberta
  - Leukemia/BMT Program of BC, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Siegel DS, Martin T, Wang M, Vij R, Jakubowiak AJ, Lonial S, Trudel S, Kukreti V, Bahlis N, Alsina M, Chanan-Khan A, Buadi F, Reu FJ, Somlo G, Zonder J, Song K, Stewart AK, Stadtmauer E, Kunkel L, Wear S, Wong AF, Orlowski RZ, Jagannath S. A phase 2 study of single-agent carfilzomib (PX-171-003-A1) in patients with relapsed and refractory multiple myeloma. Blood. 2012 Oct 4;120(14):2817-25. doi: 10.1182/blood-2012-05-425934. Epub 2012 Jul 25. PMID 22833546

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Results of this study are reported in 2 parts, depending on whether a patient was enrolled and treated under the original protocol (referred to as 'A0') or under Amendment 1 and subsequent amendments (referred to as 'A1').
Groups:
- Carfilzomib (A0): Subjects will receive carfilzomib 20 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16 of 28 day cycles
- Carfilzomib (A1): In Cycle 1, subjects will receive carfilzomib 20 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16. If all doses are administered and well-tolerated over the 28-day cycle, beginning with Cycle 2 the dose will escalate to 27 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16 for all subsequent cycles.
Period: Overall Study
Arm/Group | Carfilzomib (A0) | Carfilzomib (A1)
Started | 46 | 266
Completed | 4 (Number of patients who completed 12 cycles of treatment) | 40 (Number of patients who completed 12 cycles of treatment)
Not Completed | 42 | 226
Not completed — Adverse Event | 13 | 33
Not completed — Withdrawal by Subject | 2 | 22
Not completed — Progressive Disease | 23 | 157
Not completed — various reasons | 4 | 14

BASELINE CHARACTERISTICS:
Population: Safety population: The safety population consists of all enrolled patients who received at least 1 dose of carfilzomib.
Groups:
- Carfilzomib (A0): Subjects will receive carfilzomib 20 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16 of 28 day cycle
- Total: Total of all reporting groups
Arm/Group | Carfilzomib (A0) | Carfilzomib (A1) | Total
Number analyzed (Participants) | 46 | 266 | 312
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 146 | 172
  >=65 years | 20 | 120 | 140
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 111 | 132
  Male | 25 | 155 | 180

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (ORR)
Description: For both A0 and A1, to evaluate the best overall response rate (stringent complete response [sCR]+ complete response [CR]+ very good partial response [VGPR]+ partial response [PR]) in patients with multiple myeloma who had previously received bortezomib and either thalidomide or lenalidomide, had relapsed after two or more therapies, and were refractory to the most recently received therapy
Time Frame: A0: Subjects evaluated for disease response on Day 24 of Cycles 2, 4, 6, 9, and 12. Onset of response measured on Day 15 of Cycle 1. A1: Subjects evaluated for disease response on Day 15 of Cycle 1, Day 1 of Cycles 2 through 12 and at End of Study.
Population: Analysis population described in reporting groups below
Measure: Number (95% Confidence Interval); unit: % of participants w/ PR or better
Groups:
- Carfilzomib (A0): Subjects will receive carfilzomib 20 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16 of a 28 day cycle
  Response-evaluable Population: Enrolled patients who completed at least 1 cycle of carfilzomib and who underwent disease assessments at Screening, Cycle 1 Day 15, and Cycle 2 Day 24. This analysis set also included patients who discontinued treatment during this time due to an AE that was considered probably related to carfilzomib.
- Carfilzomib (A1): In Cycle 1, subjects will receive carfilzomib 20 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16.If all doses are administered and well-tolerated over the 28-day cycle, beginning with Cycle 2 the dose will escalate to 27 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16 for all subsequent cycles.
  Response-Evaluable Population:
  1. had measurable disease at Baseline
  2. received at least 1 dose of carfilzomib
  3. underwent baseline disease response assessments and at least 1 post-baseline disease assessment, or discontinued protocol treatment before Cycle 2 Day 1 due to an AE that was considered to be possibly or probably related to carfilzomib
Arm/Group | Carfilzomib (A0) | Carfilzomib (A1)
Number analyzed (Participants) | 42 | 257
% of participants w/ PR or better | 16.7 [6.97 to 31.36] | 23.7 [18.67 to 29.42]

2. Secondary Outcome: Clinical Benefit Response (CBR) (A0 Only)
Description: sCR, CR, VGPR, PR, and minimal response (MR)
Time Frame: Response assessments same as described in primary outcome measure
Population: Response-evaluable Population: Enrolled patients who completed at least 1 cycle of carfilzomib and who underwent disease assessments at Screening, Cycle 1 Day 15, and Cycle 2 Day 24. This analysis set also included patients who discontinued treatment during this time due to an AE that was considered probably related to carfilzomib.
Measure: Number; unit: participants
Groups:
- Carfilzomib (A0): Subjects will receive carfilzomib 20 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16 of 28 day cycle.
  Assessed by principal investigator.
Arm/Group | Carfilzomib (A0)
Number analyzed (Participants) | 42
participants
  Clinical Benefit Response (sCR+CR+VGPR+PR+MR) | 10
  Complete Response | 0
  Very Good Partial Response | 0
  Partial Response | 7
  Minimal Response | 3

3. Secondary Outcome: Clinical Benefit Response (CBR) (A1 Only)
Description: sCR, CR, VGPR, PR, and minimal response (MR)
Time Frame: Response assessments same as described in primary outcome measure
Population: Response-Evaluable Population:
  1. had measurable disease at Baseline
  2. received at least 1 dose of carfilzomib
  3. underwent baseline disease response assessments and at least 1 post-baseline disease assessment, or discontinued protocol treatment before Cycle 2 Day 1 due to an AE that was considered to be possibly or probably related to carfilzomib
Measure: Number; unit: participants
Groups:
- Carfilzomib (A1): In Cycle 1, subjects will receive carfilzomib 20 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16. If all doses are administered and well-tolerated over the 28-day cycle, beginning with Cycle 2 the dose will escalate to 27 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16 for all subsequent cycles.
  Assessed by Independent Review Committee
Arm/Group | Carfilzomib (A1)
Number analyzed (Participants) | 257
participants
  Clinical Benefit Response (sCR+CR+VGPR+PR+MR) | 95
  Complete Response | 1
  Very Good Partial Response | 13
  Partial Response | 47
  Minimal Response | 34

4. Secondary Outcome: Duration of Response (A0 Only)
Description: Duration of response (DOR) was calculated separately for subjects with clinical benefit response or overall response. DOR is defined as the time from first evidence of PR or better (for overall response) and MR or better (for clinical benefit response) to start of disease progression or death.
Time Frame: Response assessments same as described in primary outcome measure
Population: Subjects with overall response within the response-evaluable population were included in the analysis of DOR. See analysis population description of response-evaluable population above.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Carfilzomib (A0) for (ORR): Subjects will receive carfilzomib 20 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16 of a 28 day cycle
Arm/Group | Carfilzomib (A0) for (ORR)
Number analyzed (Participants) | 7
days | 219 [57 to NA] — The upper limit of the 95% confidence interval was not calculable/available (not estimable [NE]) because an insufficient number of participants reached the event at the final time point for assessment (3 of 7 responders had an event).

5. Secondary Outcome: Duration of Response (A1 Only)
Description: as for outcome 4
Time Frame: Response assessments same as described in primary outcome measure
Population: Subjects with overall response within the response-evaluable population were included in the analysis of DOR. See overall analysis population description of response-evaluable population above.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Carfilzomib (A1) for (ORR): In Cycle 1, subjects will receive carfilzomib 20 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16. If all doses are administered and well-tolerated over the 28-day cycle, beginning with Cycle 2 the dose will escalate to 27 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16 for all subsequent cycles. For subjects with ORR.
- Carfilzomib (A1) for (CBR): In Cycle 1, subjects will receive carfilzomib 20 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16. If all doses are administered and well-tolerated over the 28-day cycle, beginning with Cycle 2 the dose will escalate to 27 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16 for all subsequent cycles. For subjects with CBR.
Arm/Group | Carfilzomib (A1) for (ORR) | Carfilzomib (A1) for (CBR)
Number analyzed (Participants) | 61 | 95
months | 7.8 [5.6 to 9.2] | 8.3 [6.5 to 9.7]

6. Secondary Outcome: Time to Progression (A0 Only)
Description: Time to progression (TTP) is defined as the time from the study entry (first dose of carfilzomib) to disease progression.
Time Frame: Response assessments same as described in primary outcome measure
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Carfilzomib (A0): Subjects will receive carfilzomib 20 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16 of a 28 day cycle.
  Assesed by principal investigator.
Arm/Group | Carfilzomib (A0)
Number analyzed (Participants) | 42
months | 3.5 [2.4 to 6.7]

7. Secondary Outcome: Time to Progression (A1 Only)
Description: as for outcome 6
Time Frame: Response assessments same as described in primary outcome measure
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carfilzomib (A1)
Number analyzed (Participants) | 257
months | 3.9 [2.8 to 4.8]

8. Secondary Outcome: Progression-free Survival (A0 Only)
Description: The PFS was defined as the time from the start of treatment to progressive disease (PD) determined by PI or until death.
Time Frame: Response assessments same as described in primary outcome measure
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Carfilzomib (A0): Subjects will receive carfilzomib 20 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16 of a 28 day cycle
Arm/Group | Carfilzomib (A0)
Number analyzed (Participants) | 42
months | 3.5 [2.4 to 6.7]

9. Secondary Outcome: Progression-free Survival (A1 Only)
Description: The PFS was defined as the time from the start of treatment to progressive disease (PD) determined by PI or until death.
Time Frame: Response assessments same as described in primary outcome measure
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Carfilzomib (A1): In Cycle 1, subjects will receive carfilzomib 20 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16.If all doses are administered and well-tolerated over the 28-day cycle, beginning with Cycle 2 the dose will escalate to 27 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16 for all subsequent cycles.
Arm/Group | Carfilzomib (A1)
Number analyzed (Participants) | 257
months | 3.7 [2.8 to 4.6]

10. Secondary Outcome: Overall Survival (A1 Only)
Description: The time from start of treatment to death due to any cause OS was to be censored on the date the subject was last known to be alive for those who were alive or lost to follow-up as of a data analysis cutoff date.
Time Frame: Patients were to be followed by telephone contact for disease progression and OS every 3 months after study discontinuation for the first year and every 6 months thereafter for up to 2 years
Measure: Number (95% Confidence Interval); unit: months
Groups:
- Carfilzomib (A1) - Safety Population: In Cycle 1, subjects will receive carfilzomib 20 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16. If all doses are administered and well-tolerated over the 28-day cycle, beginning with Cycle 2 the dose will escalate to 27 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16 for all subsequent cycles.
  Safety population: The safety population was used for the analysis of safety data in this study. The safety population consists of all enrolled patients who received at least 1 dose of carfilzomib. However, for some safety analyses, at least 1 laboratory, neurological, electrocardiogram, or vital sign measurement obtained subsequent to at least 1 dose of carfilzomib was required for inclusion in the analysis of a safety specific parameter. To assess change from baseline, a baseline measurement was also required.
- Carfilzomib (A1) - Response-evaluable Population: In Cycle 1, subjects will receive carfilzomib 20 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16. If all doses are administered and well-tolerated over the 28-day cycle, beginning with Cycle 2 the dose will escalate to 27 mg/m2 intravenously on Days 1, 2, 8, 9, 15, and 16 for all subsequent cycles.
  Response-Evaluable Population(the primary analysis population) was defined as all patients who
  * had measurable disease at Baseline by either M-protein (serum and/or urine) or by quantitative serum Ig for certain patients with IgA myeloma
  * received at least 1 dose of carfilzomib
  * underwent baseline disease response assessments and at least 1 post-baseline disease assessment, or patients who discontinued protocol treatment before Cycle 2 Day 1 due to an AE that was considered to be possibly or probably related to carfilzomib-irrespective of availability of baseline and post-baseline assessment
Arm/Group | Carfilzomib (A1) - Safety Population | Carfilzomib (A1) - Response-evaluable Population
Number analyzed (Participants) | 266 | 257
months | 15.4 [12.5 to 19.0] | 15.6 [13.0 to 19.2]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) should be reported from the time the subject signs consent through 30 days post-last dose of study drug or initiation of a new anti-cancer therapy, whichever occurs first.
Arm/Group | Carfilzomib (A0) | Carfilzomib (A1)
Serious Adverse Events (participants affected / at risk) | 20/46 | 126/266
Other Adverse Events (participants affected / at risk) | 46/46 | 266/266
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib (A0) (N=46) | Carfilzomib (A1) (N=266)
Cardiac failure congestive (Cardiac disorders) | 2 | 8
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Disease progression (General disorders) | 5 | 16
Multi-organ failure (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 3
Pyrexia (General disorders) | 1 | 8
Pneumonia (Infections and infestations) | 5 | 23
Bacteraemia (Infections and infestations) | 2 | 1
Clostridium colitis (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 1 | 4
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 8
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Renal failure acute (Renal and urinary disorders) | 4 | 9
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Ventricular dysfunction (Cardiac disorders) | 0 | 1
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Infusion related reaction (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Central line infection (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Fusobacterium infection (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 5
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Hepatic enzyme abnormal (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Fluid overload (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 6
Syncope (Nervous system disorders) | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 0 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 4
Deep vein thrombosis (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib (A0) (N=46) | Carfilzomib (A1) (N=266)
Anaemia (Blood and lymphatic system disorders) | 34 | 122
Thrombocytopenia (Blood and lymphatic system disorders) | 23 | 103
Lymphopenia (Blood and lymphatic system disorders) | 16 | 62
Leukopenia (Blood and lymphatic system disorders) | 10 | 37
Neutropenia (Blood and lymphatic system disorders) | 10 | 48
Nausea (Gastrointestinal disorders) | 16 | 119
Diarrhoea (Gastrointestinal disorders) | 15 | 86
Vomiting (Gastrointestinal disorders) | 8 | 59
Constipation (Gastrointestinal disorders) | 6 | 56
Abdominal pain (Gastrointestinal disorders) | 5 | 16
Dyspepsia (Gastrointestinal disorders) | 5 | 26
Fatigue (General disorders) | 32 | 130
Pyrexia (General disorders) | 15 | 83
Asthenia (General disorders) | 7 | 40
Oedema peripheral (General disorders) | 9 | 62
Chest discomfort (General disorders) | 5 | 6
Chills (General disorders) | 5 | 42
Disease progression (General disorders) | 5 | 17
Injection site irritation (General disorders) | 4 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 17 | 71
Pneumonia (Infections and infestations) | 5 | 32
Nasopharyngitis (Infections and infestations) | 3 | 13
Blood creatinine increased (Investigations) | 16 | 67
Blood bicarbonate decreased (Investigations) | 14 | 6
Aspartate aminotransfersae increased (Investigations) | 9 | 27
Blood chloride increased (Investigations) | 8 | 1
Blood urea increased (Investigations) | 7 | 4
Blood uric acid increased (Investigations) | 7 | 15
Blood glucose increased (Investigations) | 5 | 2
Blood lactate dehydrogenase increased (Investigations) | 4 | 8
Carbon dioxide decreased (Investigations) | 4 | 2
Alanine aminotransferase decreased (Investigations) | 3 | 1
Alanine aminotransferase increased (Investigations) | 3 | 20
Insomnia (Psychiatric disorders) | 12 | 39
Confusional state (Psychiatric disorders) | 6 | 17
Renal failure acute (Renal and urinary disorders) | 4 | 13
Proteinuria (Renal and urinary disorders) | 3 | 0
Renal failure (Renal and urinary disorders) | 3 | 10
Neutrophil percentage increased (Investigations) | 3 | 0
White blood cell count decreased (Investigations) | 3 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 16 | 14
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 | 14
Anorexia (Metabolism and nutrition disorders) | 10 | 35
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 65
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 90
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 4 | 9
Hypercalcaemia (Metabolism and nutrition disorders) | 7 | 36
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 29
Hyperphosphataemia (Metabolism and nutrition disorders) | 6 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 32
Hypermagnesaemia (Metabolism and nutrition disorders) | 5 | 3
Decreased appetite (Metabolism and nutrition disorders) | 4 | 19
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 6
Chest wall pain (Musculoskeletal and connective tissue disorders) | 8 | 32
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 32
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 31
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 49
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 63
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 23
Shoulder pain (Musculoskeletal and connective tissue disorders) | 5 | 28
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 | 1
Headache (Nervous system disorders) | 12 | 74
Hypoaesthesia (Nervous system disorders) | 5 | 25
Areflexia (Nervous system disorders) | 4 | 14
Neuropathic pain (Nervous system disorders) | 4 | 9
Neuropathy peripheral (Nervous system disorders) | 4 | 17
Dizziness (Nervous system disorders) | 3 | 30
Hyporeflexia (Nervous system disorders) | 3 | 18
Neuropathy (Nervous system disorders) | 3 | 9
Paraesthesia (Nervous system disorders) | 3 | 20
Infusion site pain (General disorders) | 2 | 24
Pain (General disorders) | 2 | 24
Urinary tract infection (Infections and infestations) | 0 | 19
Contusion (Injury, poisoning and procedural complications) | 2 | 14
Weight decreased (Investigations) | 1 | 20
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 31
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 26
Dehydration (Metabolism and nutrition disorders) | 1 | 18
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 22
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 17
Anxiety (Psychiatric disorders) | 2 | 16
Depression (Psychiatric disorders) | 2 | 14
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 33
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 29
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 21
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 20
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 17
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 16
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 14
Rash (Skin and subcutaneous tissue disorders) | 3 | 20
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 17
Hypertension (Vascular disorders) | 4 | 39
Hypotension (Vascular disorders) | 4 | 21
Dry mouth (Gastrointestinal disorders) | 3 | 4
Blood albumin decreased (Investigations) | 3 | 4
Blood calcium increased (Investigations) | 3 | 5
Blood sodium decreased (Investigations) | 3 | 0
Blood phosphorus decreased (Investigations) | 3 | 12
Lymphocyte percentage decreased (Investigations) | 3 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 9 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 28
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the study is completed and all case report forms have been sent to Sponsor, Institution shall have the right to publish or otherwise make public any data resulting from the study under this agreement after publication of a multi-center publication coordinated by Sponsor with respect to the data resulting from the study, or 12 months after the Study is completed at all participating sites if a multi-center publication is not submitted by Sponsor for publication within such 12 month period.